CLINICAL TRIAL: NCT01305408
Title: A Double-Blind, Placebo-Controlled, Parallel-Group, Fixed-Dosage Study to Evaluate the Efficacy and Safety of Armodafinil Treatment (150 mg/Day) as Adjunctive Therapy in Adults With Major Depression Associated With Bipolar I Disorder
Brief Title: Study to Evaluate the Efficacy and Safety of Armodafinil Treatment (150 mg/Day) as Adjunctive Therapy in Adults With Major Depression Associated With Bipolar I Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cephalon (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C10953/3073; 2010-023623-26 (EudraCT Number)
Record Dates: First submitted 2011-02-25; First posted 2011-02-28 (Estimated); Results first posted 2015-01-26 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-04

CONDITIONS: Depression
Keywords: Bipolar I Disorder
MeSH Terms: conditions — Depression | interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Participants began taking placebo to match armodafinil and following the same titration procedure. Treatment was administered for a total of 8 weeks.
  Interventions: Drug: Placebo
- Armodafinil 150 mg/day (Experimental): Participants began taking armodafinil at a dosage of 50 mg/day; the dosage was increased by 50 mg/day on days 2 and 4, up to a dosage of 150 mg/day. Treatment was administered for a total of 8 weeks.
  Interventions: Drug: Armodafinil

INTERVENTIONS:
Drug: Armodafinil — Armodafinil tablets, taken orally, once daily in the morning
  Other Names: Nuvigil; CEP-10953
  Arms: Armodafinil 150 mg/day
Drug: Placebo — Matching placebo tablets, taken orally, once daily in the morning
  Arms: Placebo

SUMMARY:
The primary objective of the study is to determine whether armodafinil treatment, at a dosage of 150 mg/day, is more effective than placebo treatment as adjunctive therapy to mood stabilizers for treatment of adults with major depression associated with bipolar I disorder.

ELIGIBILITY:
Inclusion Criteria:

* The patient has a diagnosis of bipolar I disorder according to Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (Text Revision) (DSM-IV-TR) criteria and is currently experiencing a major depressive episode.
* Documentation that the patient has had at least 1 previous manic or mixed episode.
* The patient has had no more than 6 mood episodes in the last year.
* The patient's current major depressive episode must have started no less than 2 weeks and no more than 12 months prior to the screening visit. The current depressive episode must have begun after the patient's current mood stabilizer regime began.
* The patient must have been taking 1 (or 2) of the following protocol-allowed mood stabilizers: lithium, valproic acid, lamotrigine, aripiprazole, olanzapine, quetiapine, risperidone, ziprasidone (only if taken in combination with lithium, valproic acid, or lamotrigine). The following criteria must also be met:

  1. The mood stabilizer(s) must have been taken a minimum 4 weeks before the onset of the major depressive episode and still be taken at the time of the screening visit at dose or blood level considered appropriate for maintenance therapy by the patient's physician.
  2. The patient must continue to take the same mood stabilizer(s) during the screening period; no mood stabilizer may be added during the screening period.
  3. The mood stabilizer(s) must be taken for a minimum of at least 8 weeks prior to the baseline visit.
  4. The dosage of the mood stabilizer(s) must be stable for a minimum of 4 weeks prior to the baseline visit.
  5. The mood stabilizer(s) must be taken in an oral formulation, with the exception of risperidone, which can be either in an oral or long-acting injection formulation.
  6. The patient may be taking 2 protocol-allowed mood stabilizers only if 1 of the drugs is lithium, valproic acid, or lamotrigine.

Exclusion Criteria:

* The patient has any Axis I disorder apart from bipolar I disorder that was the primary focus of treatment within 6 months of the screening visit or during the screening period.
* The patient has psychotic symptoms or has had psychosis within 4 weeks of the screening visit or during the screening period.
* The patient has current active suicidal ideation, is at imminent risk of self-harm, or has a history of significant suicidal ideation or suicide attempt at any time in the past that causes concern at present.
* The patient has a history of an eating disorder or obsessive compulsive disorder (OCD) within 6 months of the screening visit or during the screening period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 399 (Actual)
Dates: Start 2011-03; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sponsor's Medical Expert, Study Director — Cephalon
Locations (130):
- United States (28):
  - Teva Investigational Site 225, Birmingham, Alabama
  - Teva Investigational Site 295, Sherman Oaks, California
  - Teva Investigational Site 122, Temecula, California
  - Teva Investigational Site 606, Jacksonville Beach, Florida
  - Teva Investigational Site 127, Lauderhill, Florida
  - Teva Investigational Site 608, Tampa, Florida
  - Teva Investigational Site 116, Atlanta, Georgia
  - Teva Investigational Site 205, Atlanta, Georgia
  - Teva Investigational Site 195, Park Ridge, Illinois
  - Teva Investigational Site 611, Indianapolis, Indiana
  - Teva Investigational Site 600, Lafayette, Indiana
  - Teva Investigational Site 603, Watertown, Massachusetts
  - Teva Investigational Site 207, Brooklyn, New York
  - Teva Investigational Site 202, New York, New York
  - Teva Investigational Site 110, Staten Island, New York
  - Teva Investigational Site 411, Staten Island, New York
  - Teva Investigational Site 614, Wilmington, North Carolina
  - Teva Investigational Site 610, Cincinnati, Ohio
  - Teva Investigational Site 615, Toledo, Ohio
  - Teva Investigational Site 401, Oklahoma City, Oklahoma
  - Teva Investigational Site 609, Oklahoma City, Oklahoma
  - Teva Investigational Site 616, Oklahoma City, Oklahoma
  - Teva Investigational Site 406, Allentown, Pennsylvania
  - Teva Investigational Site 403, DeSoto, Texas
  - Teva Investigational Site 612, Friendswood, Texas
  - Teva Investigational Site 408, Salt Lake City, Utah
  - Teva Investigational Site 613, Kirkland, Washington
  - Teva Investigational Site 605, Spokane, Washington
- Argentina (15):
  - Teva Investigational Site 134, Buenos Aires
  - Teva Investigational Site 136, Buenos Aires
  - Teva Investigational Site 881, Buenos Aires
  - Teva Investigational Site 884, Buenos Aires
  - Teva Investigational Site 888, Buenos Aires
  - Teva Investigational Site 236, Córdoba
  - Teva Investigational Site 135, Córdoba Capital
  - Teva Investigational Site 371, La Plata
  - Teva Investigational Site 886, La Plata
  - Teva Investigational Site 138, La Plata, Buenos Aires
  - Teva Investigational Site 882, Mendoza
  - Teva Investigational Site 883, Mendoza
  - Teva Investigational Site 885, Mendoza
  - Teva Investigational Site 887, Mendoza
  - Teva Investigational Site 238, Rosario
- Brazil (7):
  - Teva Investigational Site 623, Belo Horizonte
  - Teva Investigational Site 626, Curitiba-Parana
  - Teva Investigational Site 621, Distrito de Rubiao Junior
  - Teva Investigational Site 627, Itapira -Sao Paulo
  - Teva Investigational Site 624, Rio de Janeiro
  - Teva Investigational Site 622, Salvador
  - Teva Investigational Site 628, São Paulo
- Bulgaria (16):
  - Teva Investigational Site 248, Burgas
  - Teva Investigational Site 146, Kardzhali
  - Teva Investigational Site 148, Kazanlak
  - Teva Investigational Site 853, Pazardzhik
  - Teva Investigational Site 852, Pleven
  - Teva Investigational Site 145, Plovdiv
  - Teva Investigational Site 370, Rousse
  - Teva Investigational Site 147, Sofia
  - Teva Investigational Site 149, Sofia
  - Teva Investigational Site 244, Sofia
  - Teva Investigational Site 247, Sofia
  - Teva Investigational Site 854, Sofia
  - Teva Investigational Site 855, Sofia
  - Teva Investigational Site 245, Varna
  - Teva Investigational Site 851, Varna
  - Teva Investigational Site 856, Varna
- Croatia (5):
  - Teva Investigational Site 635, Rijeka
  - Teva Investigational Site 631, Split
  - Teva Investigational Site 632, Zagreb
  - Teva Investigational Site 633, Zagreb
  - Teva Investigational Site 634, Zagreb
- Finland (4):
  - Teva Investigational Site 716, Helsinki
  - Teva Investigational Site 717, Helsinki
  - Teva Investigational Site 719, Kangasala
  - Teva Investigational Site 718, Turku
- Germany (6):
  - Teva Investigational Site 655, Achim
  - Teva Investigational Site 656, Berlin
  - Teva Investigational Site 653, Cologne
  - Teva Investigational Site 651, Dresden
  - Teva Investigational Site 654, Freiburg im Breisgau
  - Teva Investigational Site 652, Mittweida
- Hungary (5):
  - Teva Investigational Site 661, Budapest
  - Teva Investigational Site 662, Budapest
  - Teva Investigational Site 664, Budapest
  - Teva Investigational Site 665, Győr
  - Teva Investigational Site 666, Nagykálló
- Italy (8):
  - Teva Investigational Site 688, Catania
  - Teva Investigational Site 689, Florence
  - Teva Investigational Site 686, Genova
  - Teva Investigational Site 691, Lido Di Camaiore(LU)
  - Teva Investigational Site 690, Naples
  - Teva Investigational Site 687, Pisa
  - Teva Investigational Site 693, Pisa
  - Teva Investigational Site 692, Roma
- Poland (7):
  - Teva Investigational Site 259, Bialystok
  - Teva Investigational Site 257, Gdansk
  - Teva Investigational Site 258, Gdynia
  - Teva Investigational Site 155, Krakow
  - Teva Investigational Site 255, Skorzewo
  - Teva Investigational Site 861, Szczecin
  - Teva Investigational Site 157, Tuszyn
- Serbia (7):
  - Teva Investigational Site 177, Belgrade
  - Teva Investigational Site 831, Belgrade
  - Teva Investigational Site 832, Belgrade
  - Teva Investigational Site 835, Belgrade
  - Teva Investigational Site 176, Kragujevac
  - Teva Investigational Site 837, Niš
  - Teva Investigational Site 834, Novi Kneževac
- Slovakia (5):
  - Teva Investigational Site 700, Bojnice
  - Teva Investigational Site 699, Bratislava
  - Teva Investigational Site 697, Rimavská Sobota
  - Teva Investigational Site 696, Rožňava
  - Teva Investigational Site 698, Trenčín
- South Africa (7):
  - Teva Investigational Site 707, Cape Town
  - Teva Investigational Site 709, Cape Town
  - Teva Investigational Site 712, Cape Town
  - Teva Investigational Site 708, Centurion
  - Teva Investigational Site 710, Johannesburg
  - Teva Investigational Site 711, Paarl
  - Teva Investigational Site 706, Pretoria
- Ukraine (10):
  - Teva Investigational Site 181, Dnipropetrovsk
  - Teva Investigational Site 872, Donetsk
  - Teva Investigational Site 282, Kharkiv
  - Teva Investigational Site 281, Kiev
  - Teva Investigational Site 180, Luhansk
  - Teva Investigational Site 873, Lviv
  - Teva Investigational Site 875, Odesa
  - Teva Investigational Site 183, Poltava
  - Teva Investigational Site 871, S. Oleksandrivka
  - Teva Investigational Site 182, Vinnytsia

REFERENCES:
- [Derived] Frye MA, Amchin J, Bauer M, Adler C, Yang R, Ketter TA. Randomized, placebo-controlled, adjunctive study of armodafinil for bipolar I depression: implications of novel drug design and heterogeneity of concurrent bipolar maintenance treatments. Int J Bipolar Disord. 2015 Dec;3(1):34. doi: 10.1186/s40345-015-0034-0. Epub 2015 Sep 2. PMID 26330288

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Region 1: USA and Canada Region 2: Eastern European countries, Kyrgyzstan, Mongolia, Uzbekistan, Cyprus, Greece, and Turkey Region 3: Central and Northern European countries, Andorra, Australia, Iceland, Monaco, San Marino, and Vatican City Region 4: Rest of World
Pre-assignment Details: Participants were randomized (1:1) to receive150 mg/day armodafinil or matching placebo. Randomization was stratified on the basis of the mood-stabilizing medication and region of the world.
Period: Overall Study
Arm/Group | Placebo | Armodafinil 150 mg/Day
Started | 199 | 200
Safety Population | 198 (Treated participants. One participant was randomized but not treated.) | 200 (Treated participants.)
Full Analysis Population | 196 (Treated participants who have at least 1 postbaseline IDS-C30 efficacy assessment) | 197 (Treated participants who have at least 1 postbaseline IDS-C30 efficacy assessment)
Completed | 167 | 169
Not Completed | 32 | 31
Not completed — Adverse Event | 10 | 7
Not completed — Lack of Efficacy | 3 | 4
Not completed — Withdrawal by Subject | 9 | 9
Not completed — Protocol Violation | 4 | 6
Not completed — Lost to Follow-up | 5 | 3
Not completed — Noncompliance with study medication | 0 | 1
Not completed — Noncompliance with study procedures | 0 | 1
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Population: Randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Armodafinil 150 mg/Day | Total
Number analyzed (Participants) | 199 | 200 | 399
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.7 (11.62) | 45.3 (11.26) | 44.5 (11.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 121 | 120 | 241
  Male | 78 | 80 | 158
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 22 | 36
  Not Hispanic or Latino | 183 | 176 | 359
  Unknown or Not Reported | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 16 | 14 | 30
  White | 176 | 182 | 358
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 0 | 6
Weight [Mean (Standard Deviation); unit: kg] | 81.2 (17.46) | 80.7 (17.54) | 80.9 (17.48)
Height [Mean (Standard Deviation); unit: cm] | 168.4 (9.32) | 168.9 (9.23) | 168.6 (9.27)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 28.7 (5.95) | 28.2 (5.52) | 28.4 (5.73)
Time Since Start of Current Depressive Episode [Mean (Standard Deviation); unit: weeks] | 12.1 (9.10) | 12.3 (9.89) | 12.2 (9.49)
Time Since First Diagnosis for Bipolar [Mean (Standard Deviation); unit: years] | 9.9 (8.72) | 10.7 (8.55) | 10.3 (8.63)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 8 in the Total Score From the 30-Item Inventory of Depressive Symptomatology-Clinician-Rated (IDS-C30)
Description: The IDS-C30 is a standardized 30-item, clinician-rated scale to assess the severity of a participant's depressive symptoms. Every effort was made to have the same rater evaluate a participant across all visits.
  Total scores range from 0-84, with a score of 0 indicating no depression and a score of 84 indicating the most severe depression. Negative change from baseline values indicate improvement in the severity of depression.
Time Frame: Day 0 (baseline), Week 8
Population: Full analysis set which includes participants who took 1 or more doses of study drug and who have at least 1 postbaseline IDS-C30 efficacy assessment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Armodafinil 150 mg/Day
Number analyzed (Participants) | 196 | 197
units on a scale | -19.4 (0.99) | -20.8 (0.99)
Statistical Analysis 1: Comparison: Placebo vs Armodafinil 150 mg/Day; Test type: Superiority or Other; p = 0.2717, mixed-model repeated measures (MMRM) — Statistical tests were 2-tailed at the 0.05 level of significance; Treatment, visit, treatment-by-visit interaction, concurrent mood-stabilizing medication, and region of the world used as fixed factors; Mean Difference (Final Values) = -1.4, 95% CI 2-sided [-3.76 to 1.06]

2. Secondary Outcome: Percentage of Responders At Different Treatment Weeks According to the 30-Item Inventory of Depressive Symptomatology-Clinician Rated (IDS-C30) Total Score
Description: A responder is a participant with a ≥50% decrease or greater from baseline in the total score of the IDS-C30. The IDS-C30 is a standardized 30-item, clinician-rated scale to assess the severity of a participant's depressive symptoms. Every effort was made to have the same rater evaluate a participant across all visits.
  Total scores range from 0-84, with a score of 0 indicating no depression and a score of 84 indicating the most severe depression.
Time Frame: Day 0 (baseline), Weeks 1, 2, 4, 6, 7, and 8, and last postbaseline observation (up to 8 weeks)
Population: Full analysis set which includes participants who took 1 or more doses of study drug and who have at least 1 postbaseline IDS-C30 efficacy assessment. The denominator for calculating the percentages at each visit is the number of participants with a nonmissing value at that visit. Endpoint was the last observed postbaseline data.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Armodafinil 150 mg/Day
Number analyzed (Participants) | 196 | 197
percentage of participants
  Week 1 (196, 195) | 2 | 3
  Week 2 (187, 189) | 13 | 9
  Week 4 (181, 183) | 21 | 27
  Week 6 (172, 172) | 29 | 41
  Week 7 (167, 170) | 39 | 51
  Week 8 (167, 169) | 46 | 56
  Endpoint (196, 197) | 41 | 49

3. Secondary Outcome: Percentage of Participants in Remission At Different Treatment Weeks According to the 30-Item Inventory of Depressive Symptomatology-Clinician Rated (IDS-C30) Total Score
Description: A participant in remission was defined as a participant with an IDS-C30 total score of 11 or less.
  The IDS-C30 is a standardized 30-item, clinician-rated scale to assess the severity of a participant's depressive symptoms. Every effort was made to have the same rater evaluate a participant across all visits.
  Total scores range from 0-84, with a score of 0 indicating no depression and a score of 84 indicating the most severe depression.
Time Frame: Weeks 1, 2, 4, 6, 7, and 8, and last postbaseline observation (up to 8 weeks)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Armodafinil 150 mg/Day
Number analyzed (Participants) | 196 | 197
percentage of participants
  Week 1 (196, 195) | .5 | 1
  Week 2 (187, 189) | 2 | 2
  Week 4 (181, 183) | 5 | 7
  Week 6 (172, 172) | 9 | 12
  Week 7 (167, 170) | 14 | 19
  Week 8 (167, 169) | 15 | 26
  Endpoint (196, 197) | 13 | 22

4. Secondary Outcome: Change From Baseline to Different Treatment Weeks in the Total Score From the 30-Item Inventory of Depressive Symptomatology-Clinician-Rated (IDS-C30)
Description: as for outcome 1
Time Frame: Day 0 (baseline), Weeks 1, 2, 4, 6, 7, and 8, and last postbaseline observation (up to 8 weeks)
Population: Full analysis set which includes participants who took 1 or more doses of study drug and who have at least 1 postbaseline IDS-C30 efficacy assessment. Participants are included in the analysis at each timepoint if they have a nonmissing value at that visit. Endpoint for analyses was the last observed postbaseline data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Armodafinil 150 mg/Day
Number analyzed (Participants) | 196 | 197
units on a scale
  Week 1 (196, 195) | -6.0 (6.61) | -5.3 (7.12)
  Week 2 (187, 189) | -10.0 (8.71) | -8.9 (8.56)
  Week 4 (181, 183) | -13.4 (9.87) | -13.5 (10.54)
  Week 6 (172, 172) | -15.8 (10.42) | -17.6 (11.09)
  Week 7 (167, 170) | -18.0 (11.42) | -20.2 (10.88)
  Week 8 (167, 169) | -19.7 (11.30) | -21.6 (11.75)
  Endpoint (196, 197) | -18.3 (11.62) | -19.5 (12.66)

5. Secondary Outcome: Change From Baseline to Different Treatment Weeks in the Total Score From the 16-Item Quick Inventory of Depressive Symptomatology-Clinician-Rated (QIDS-C16)
Description: The QIDS-C16 was derived from specified items in the IDS-C30, clinician-rated scale to assess the severity of a participant's depressive symptoms. Total scores range from 0-27, with a score of 0 indicating no depression and a score of 27 indicating the most severe depression. Negative change from baseline values indicate improvement in the severity of depression.
Time Frame: Day 0 (baseline), Weeks 1, 2, 4, 6, 7, and 8, and last postbaseline observation (up to 8 weeks)
Population: Full analysis set which includes participants who took 1 or more doses of study drug and who have at least 1 postbaseline IDS-C30 efficacy assessment. The number of participants at each visit are those with a nonmissing value at that visit. Endpoint was the last observed postbaseline data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Armodafinil 150 mg/Day
Number analyzed (Participants) | 196 | 197
units on a scale
  Week 1 (196, 195) | -2.4 (2.92) | -2.1 (3.07)
  Week 2 (187, 189) | -4.2 (3.83) | -3.4 (3.63)
  Week 4 (181, 183) | -5.3 (4.05) | -5.3 (4.15)
  Week 6 (172, 172) | -6.3 (4.16) | -6.7 (4.38)
  Week 7 (167, 170) | -7.2 (4.49) | -7.8 (4.35)
  Week 8 (167, 169) | -8.0 (4.53) | -8.3 (4.62)
  Endpoint (196, 197) | -7.3 (4.73) | -7.5 (4.91)

6. Secondary Outcome: Change From Baseline to Different Treatment Weeks in the Clinical Global Impression of Severity (CGI-S) for Depression
Description: The CGI-S is an observer-rated scale that measures illness severity on a 7-point scale, with the severity of illness scale using a range of responses from 1 (normal) through to 7 (amongst the most severely ill patients). Negative change from baseline values indicate improvement in the severity of depression.
Time Frame: Day 0 (baseline), Weeks 1, 2, 4, 6, 7, and 8, and last postbaseline observation (up to 8 weeks)
Population: Full analysis set which includes participants who took 1 or more doses of study drug and who have at least 1 postbaseline IDS-C30 efficacy assessment. The number of participants is those with a nonmissing value at that visit. Endpoint was the last observed postbaseline data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Armodafinil 150 mg/Day
Number analyzed (Participants) | 196 | 197
units on a scale
  Week 1 (196, 195) | -0.2 (0.49) | -0.2 (0.46)
  Week 2 (187, 189) | -0.5 (0.65) | -0.5 (0.77)
  Week 4 (181, 183) | -0.7 (0.76) | -0.9 (0.97)
  Week 6 (172, 172) | -1.0 (0.91) | -1.2 (1.03)
  Week 7 (167, 170) | -1.2 (1.08) | -1.4 (1.10)
  Week 8 (167, 169) | -1.3 (1.11) | -1.6 (1.19)
  Endpoint (196, 197) | -1.2 (1.14) | -1.4 (1.25)

7. Secondary Outcome: Change From Baseline to Weeks 4, 8 and Endpoint in the Global Assessment for Functioning (GAF) Scale
Description: The Global Assessment of Functioning (GAF) is a numeric scale (1 through 100) used by mental health clinicians and physicians to rate subjectively the social, occupational, and psychological functioning of adults, e.g., how well or adaptively one is meeting various problems-in-living. Ratings of 1 - 10 mean the participant is in persistent danger of severely hurting self or others (e.g., recurrent violence) or persistent inability to maintain minimal personal hygiene or serious suicidal act with clear expectation of death. Ratings of 91 - 100 indicate no symptoms, and the participant exhibits superior functioning in a wide range of activities, life's problems never seem to get out of hand, is sought out by others because of his or her many positive qualities. Positive change from baseline values indicate improvement in functioning.
Time Frame: Day 0 (baseline), Weeks 4, 8, and last postbaseline observation (up to 8 weeks)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Armodafinil 150 mg/Day
Number analyzed (Participants) | 196 | 197
units on a scale
  Week 4 (181, 183) | 5.8 (7.39) | 8.2 (10.39)
  Week 8 (167, 169) | 11.5 (10.42) | 15.3 (11.72)
  Endpoint (189, 192) | 10.6 (10.42) | 13.6 (12.38)

8. Secondary Outcome: Participants With Treatment-Emergent Adverse Events (TEAE)
Description: AEs were graded by the investigator for severity on a three-point scale: mild, moderate and severe. Causality is graded as either related or not related. A serious adverse event (SAE) is an AE resulting in death, a life-threatening adverse event, hospitalization, a persistent or significant disability/incapacity, a congenital anomaly/birth defect, or an important medical event that may require medical intervention to prevent any of the previous results.
  Protocol-defined adverse events requiring expedited reporting included skin rash, hypersensitivity reaction, emergent suicidal ideation or suicide attempt, and psychosis.
Time Frame: Day 1 to Week 9
Population: The safety analysis set includes randomized participants who took 1 or more doses of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | Armodafinil 150 mg/Day
Number analyzed (Participants) | 198 | 200
participants
  >=1 adverse event | 71 | 89
  Severe adverse event | 4 | 4
  Treatment-related adverse event | 32 | 53
  Deaths | 0 | 0
  Other serious adverse events | 6 | 5
  Withdrawn from study due to adverse events | 10 | 7
  Protocol-defined adverse events | 3 | 3

9. Secondary Outcome: Change From Baseline to Endpoint in the Young Mania Rating Scale (YMRS) Total Score
Description: The YMRS is a clinician-rated, 11-item checklist used to measure the severity of manic episodes. Information for assigning scores is gained from the participant's subjective reported symptoms over the previous 48 hours and from clinical observation during the interview. Seven items are ranked 0 through 4 and have descriptors associated with each severity level. Four items (irritability, speech, content, and disruptive-aggressive behavior) are scored 0 through 8 and have descriptors for every second increment. The total scale is 0-60. A score of ≤12 indicates remission of manic symptoms, and higher scores indicate greater severity of mania. Negative change from baseline scores indicate a decrease in severity of mania.
Time Frame: Day 0 (baseline), last postbaseline observation (up to 8 weeks)
Population: The safety analysis set includes randomized participants who took 1 or more doses of study drug. The number analyzed includes participants with both baseline and during treatment assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Armodafinil 150 mg/Day
Number analyzed (Participants) | 196 | 198
units on a scale | -1.0 (2.45) | -0.9 (3.19)

10. Secondary Outcome: Change From Baseline to Endpoint in the Hamilton Anxiety Scale (HAM-A) Total Score
Description: HAM-A measures the severity of anxiety symptoms. The scale consists of 14 items, each defined by a series of symptoms, and measures both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety). Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe. Negative change from baseline scores indicate a decrease in severity of anxiety.
Time Frame: Day 0 (baseline), last postbaseline observation (up to 8 weeks)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Armodafinil 150 mg/Day
Number analyzed (Participants) | 190 | 194
units on a scale | -4.2 (4.53) | -4.3 (5.37)

11. Secondary Outcome: Change From Baseline to Endpoint in the Insomnia Severity Index (ISI) Total Score
Description: The ISI is a participant-rated, 7-item questionnaire designed to assess the severity of the participant's insomnia. Each item is ranked 0 (none) through 4 (very severe) and has a descriptor associated with each severity level. Total range is 0 (no insomnia) to 28 (very severe insomnia). Responses to each item are added to obtain a total score to determine the severity of insomnia. Negative change from baseline scores indicate a decrease in severity of insomnia.
Time Frame: Day 0 (baseline), last postbaseline observation (up to 8 weeks)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Armodafinil 150 mg/Day
Number analyzed (Participants) | 190 | 192
units on a scale | -7.0 (6.62) | -7.1 (6.91)

12. Secondary Outcome: Columbia-Suicide Severity Rating Scale 'Since Last Visit' Version (C-SSRS-SLV) For Weeks 1, 2, 4, 6, 7, 8, and Endpoint For the Suicidal Behavior - Actual Attempt Question
Description: The C-SSRS is a clinician-rated scale that assesses suicidality from ideation to behaviors and monitors the potential emergence of suicidality in clinical studies. The C-SSRS-B (baseline) was performed at screening and the C-SSRS-SLV ('Since Last Visit') was performed at baseline and weeks 1, 2, 4, 6, 7, and 8 or last postbaseline observation. The Suicidal Behavior - Actual Attempt question records whether the participant committed a potentially self-injurious act with at least some wish to die since the last visit.
Time Frame: Weeks 1, 2, 4, 6, 7, and 8, and last postbaseline observation (up to 8 weeks)
Population: The safety analysis set includes randomized participants who took 1 or more doses of study drug. The number analyzed includes participants with treatment assessments at the indicated time period.
Measure: Number; unit: participants
Arm/Group | Placebo | Armodafinil 150 mg/Day
Number analyzed (Participants) | 198 | 200
participants
  Week 1 (196, 195) | 0 | 0
  Week 2 (187, 189) | 0 | 0
  Week 4 (181, 183) | 0 | 0
  Week 6 (172, 172) | 0 | 0
  Week 7 (167, 170) | 0 | 0
  Week 8 (167, 169) | 0 | 0
  Endpoint (196, 198) | 0 | 0

13. Secondary Outcome: Columbia-Suicide Severity Rating Scale 'Since Last Visit' Version (C-SSRS-SLV) For Weeks 1, 2, 4, 6, 7, 8, and Endpoint For the Suicidal Behavior - Non-Suicidal Self-Injurious Behavior Question
Description: The C-SSRS is a clinician-rated scale that assesses suicidality from ideation to behaviors and monitors the potential emergence of suicidality in clinical studies. The C-SSRS-B (baseline) was performed at screening and the C-SSRS-SLV ('Since Last Visit') was performed at baseline and weeks 1, 2, 4, 6, 7, and 8 or last postbaseline observation.
  The Suicidal Behavior - Non-Suicidal Self-Injurious Behavior question records whether the participant committed a potentially self-injurious act that was not associated with a wish to die since the last visit.
Time Frame: Weeks 1, 2, 4, 6, 7, and 8, and last postbaseline observation (up to 8 weeks)
Population: as for outcome 12
Measure: Number; unit: participants
Arm/Group | Placebo | Armodafinil 150 mg/Day
Number analyzed (Participants) | 198 | 200
participants
  Week 1 (196, 195) | 0 | 0
  Week 2 (187, 189) | 0 | 0
  Week 4 (181, 183) | 0 | 0
  Week 6 (172, 172) | 0 | 0
  Week 7 (167, 170) | 0 | 0
  Week 8 (167, 169) | 0 | 0
  Endpoint (196, 198) | 0 | 0

14. Secondary Outcome: Columbia-Suicide Severity Rating Scale 'Since Last Visit' Version (C-SSRS-SLV) For Weeks 1, 2, 4, 6, 7, 8, and Endpoint For the Suicidal Behavior - Interrupted Attempt Question
Description: The C-SSRS is a clinician-rated scale that assesses suicidality from ideation to behaviors and monitors the potential emergence of suicidality in clinical studies. The C-SSRS-B (baseline) was performed at screening and the C-SSRS-SLV ('Since Last Visit') was performed at baseline and weeks 1, 2, 4, 6, 7, and 8 or last postbaseline observation.
  The Suicidal Behavior - Interrupted Attempt question records whether the participant was interrupted by an outside circumstance from starting the potentially self-injurious act with at least some wish to die since the last visit.
Time Frame: Weeks 1, 2, 4, 6, 7, and 8, and last postbaseline observation (up to 8 weeks)
Population: as for outcome 12
Measure: Number; unit: participants
Arm/Group | Placebo | Armodafinil 150 mg/Day
Number analyzed (Participants) | 198 | 200
participants
  Week 1 (196, 195) | 0 | 0
  Week 2 (187, 189) | 0 | 0
  Week 4 (181, 183) | 0 | 0
  Week 6 (172, 172) | 0 | 0
  Week 7 (167, 170) | 0 | 0
  Week 8 (167, 169) | 0 | 0
  Endpoint (196, 198) | 0 | 0

15. Secondary Outcome: Columbia-Suicide Severity Rating Scale 'Since Last Visit' Version (C-SSRS-SLV) For Weeks 1, 2, 4, 6, 7, 8, and Endpoint For the Suicidal Behavior - Aborted Attempt Question
Description: The C-SSRS is a clinician-rated scale that assesses suicidality from ideation to behaviors and monitors the potential emergence of suicidality in clinical studies. The C-SSRS-B (baseline) was performed at screening and the C-SSRS-SLV ('Since Last Visit') was performed at baseline and weeks 1, 2, 4, 6, 7, and 8 or last postbaseline observation.
  The Suicidal Behavior - Aborted Attempt question records whether the participant began to take steps toward making a suicide attempt but stops themselves before starting the potentially self-injurious act since the last visit.
Time Frame: Weeks 1, 2, 4, 6, 7, and 8, and last postbaseline observation (up to 8 weeks)
Population: as for outcome 12
Measure: Number; unit: participants
Arm/Group | Placebo | Armodafinil 150 mg/Day
Number analyzed (Participants) | 198 | 200
participants
  Week 1 (196, 195) | 0 | 0
  Week 2 (187, 189) | 0 | 0
  Week 4 (181, 183) | 0 | 0
  Week 6 (172, 172) | 0 | 0
  Week 7 (167, 170) | 0 | 0
  Week 8 (167, 169) | 0 | 0
  Endpoint (196, 198) | 0 | 0

16. Secondary Outcome: Columbia-Suicide Severity Rating Scale 'Since Last Visit' Version (C-SSRS-SLV) For Weeks 1, 2, 4, 6, 7, 8, and Endpoint For the Suicidal Behavior - Suicidal Behavior Question
Description: The C-SSRS is a clinician-rated scale that assesses suicidality from ideation to behaviors and monitors the potential emergence of suicidality in clinical studies. The C-SSRS-B (baseline) was performed at screening and the C-SSRS-SLV ('Since Last Visit') was performed at baseline and weeks 1, 2, 4, 6, 7, and 8 or last postbaseline observation.
  The Suicidal Behavior - Suicidal Behavior question records whether in the clinician's opinion, the participant exhibited suicidal behavior since the last visit.
Time Frame: Weeks 1, 2, 4, 6, 7, and 8, and last postbaseline observation (up to 8 weeks)
Population: as for outcome 12
Measure: Number; unit: participants
Arm/Group | Placebo | Armodafinil 150 mg/Day
Number analyzed (Participants) | 198 | 200
participants
  Week 1 (196, 195) | 0 | 0
  Week 2 (187, 189) | 0 | 0
  Week 4 (181, 183) | 0 | 0
  Week 6 (172, 172) | 0 | 0
  Week 7 (167, 170) | 0 | 0
  Week 8 (167, 169) | 0 | 0
  Endpoint (196, 198) | 0 | 0

17. Secondary Outcome: Columbia-Suicide Severity Rating Scale 'Since Last Visit' Version (C-SSRS-SLV) For Weeks 1, 2, 4, 6, 7, 8, and Endpoint For the Suicidal Behavior - Preparatory Acts or Behavior Question
Description: The C-SSRS is a clinician-rated scale that assesses suicidality from ideation to behaviors and monitors the potential emergence of suicidality in clinical studies. The C-SSRS-B (baseline) was performed at screening and the C-SSRS-SLV ('Since Last Visit') was performed at baseline and weeks 1, 2, 4, 6, 7, and 8 or last postbaseline observation.
  The Suicidal Behavior - Preparatory Acts or Behavior question records whether the participant exhibited acts or preparations towards imminently making a suicide attempt since the last visit.
Time Frame: Weeks 1, 2, 4, 6, 7, and 8, and last postbaseline observation (up to 8 weeks)
Population: as for outcome 12
Measure: Number; unit: participants
Arm/Group | Placebo | Armodafinil 150 mg/Day
Number analyzed (Participants) | 198 | 200
participants
  Week 1 (196, 195) | 0 | 0
  Week 2 (187, 189) | 0 | 0
  Week 4 (181, 183) | 0 | 0
  Week 6 (172, 172) | 0 | 0
  Week 7 (167, 170) | 0 | 0
  Week 8 (167, 169) | 0 | 0
  Endpoint (196, 198) | 0 | 0

18. Secondary Outcome: Columbia-Suicide Severity Rating Scale 'Since Last Visit' Version (C-SSRS-SLV) For Weeks 1, 2, 4, 6, 7, 8, and Endpoint For the Suicidal Behavior - Completed Suicide Question
Description: The C-SSRS is a clinician-rated scale that assesses suicidality from ideation to behaviors and monitors the potential emergence of suicidality in clinical studies. The C-SSRS-B (baseline) was performed at screening and the C-SSRS-SLV ('Since Last Visit') was performed at baseline and weeks 1, 2, 4, 6, 7, and 8 or last postbaseline observation.
  The Suicidal Behavior - Completed Suicide question records whether the participant intentionally causing his/her's own death since the last visit.
Time Frame: Weeks 1, 2, 4, 6, 7, and 8, and last postbaseline observation (up to 8 weeks)
Population: as for outcome 12
Measure: Number; unit: participants
Arm/Group | Placebo | Armodafinil 150 mg/Day
Number analyzed (Participants) | 198 | 200
participants
  Week 1 (196, 195) | 0 | 0
  Week 2 (187, 189) | 0 | 0
  Week 4 (181, 183) | 0 | 0
  Week 6 (172, 172) | 0 | 0
  Week 7 (167, 170) | 0 | 0
  Week 8 (167, 169) | 0 | 0
  Endpoint (196, 198) | 0 | 0

19. Secondary Outcome: Columbia-Suicide Severity Rating Scale 'Since Last Visit' Version (C-SSRS-SLV) For Weeks 1, 2, 4, 6, 7, 8, and Endpoint For the Suicidal Ideation - Wish to Be Dead Question
Description: The C-SSRS is a clinician-rated scale that assesses suicidality from ideation to behaviors and monitors the potential emergence of suicidality in clinical studies. The C-SSRS-B (baseline) was performed at screening and the C-SSRS-SLV ('Since Last Visit') was performed at baseline and weeks 1, 2, 4, 6, 7, and 8 or last postbaseline observation.
  The Suicidal Ideation - Wish to Be Dead question records whether the participant endorses thoughts about a wish to dead or not alive anymore, or a wish to fall asleep and not wake up since the last visit.
Time Frame: Weeks 1, 2, 4, 6, 7, and 8, and last postbaseline observation (up to 8 weeks)
Population: as for outcome 12
Measure: Number; unit: participants
Arm/Group | Placebo | Armodafinil 150 mg/Day
Number analyzed (Participants) | 198 | 200
participants
  Week 1 (196, 195) | 6 | 5
  Week 2 (187, 189) | 2 | 6
  Week 4 (181, 183) | 1 | 7
  Week 6 (172, 172) | 2 | 3
  Week 7 (167, 170) | 2 | 2
  Week 8 (167, 169) | 1 | 3
  Endpoint (196, 198) | 2 | 4

20. Secondary Outcome: Columbia-Suicide Severity Rating Scale 'Since Last Visit' Version (C-SSRS-SLV) For Weeks 1, 2, 4, 6, 7, 8, and Endpoint For the Suicidal Ideation - Non-Specific Active Suicidal Thoughts Question
Description: The C-SSRS is a clinician-rated scale that assesses suicidality from ideation to behaviors and monitors the potential emergence of suicidality in clinical studies. The C-SSRS-B (baseline) was performed at screening and the C-SSRS-SLV ('Since Last Visit') was performed at baseline and weeks 1, 2, 4, 6, 7, and 8 or last postbaseline observation.
  The Suicidal Ideation - Non-Specific Active Suicidal Thoughts question records whether the participant shares general non-specific thoughts of wanting to end one's life/commit suicide since the last visit.
Time Frame: Weeks 1, 2, 4, 6, 7, and 8, and last postbaseline observation (up to 8 weeks)
Population: as for outcome 12
Measure: Number; unit: participants
Arm/Group | Placebo | Armodafinil 150 mg/Day
Number analyzed (Participants) | 198 | 200
participants
  Week 1 (196, 195) | 2 | 0
  Week 2 (187, 189) | 0 | 0
  Week 4 (181, 183) | 0 | 1
  Week 6 (172, 172) | 0 | 1
  Week 7 (167, 170) | 0 | 1
  Week 8 (167, 169) | 0 | 1
  Endpoint (196, 198) | 0 | 1

21. Secondary Outcome: Columbia-Suicide Severity Rating Scale 'Since Last Visit' Version (C-SSRS-SLV) For Weeks 1, 2, 4, 6, 7, 8, and Endpoint For the Suicidal Ideation - Any Methods (Not Plan) Without Intent to Act Question
Description: The C-SSRS is a clinician-rated scale that assesses suicidality from ideation to behaviors and monitors the potential emergence of suicidality in clinical studies. The C-SSRS-B (baseline) was performed at screening and the C-SSRS-SLV ('Since Last Visit') was performed at baseline and weeks 1, 2, 4, 6, 7, and 8 or last postbaseline observation.
  The Suicidal Ideation - Any Methods (Not Plan) Without Intent to Act question records whether the participant endorses thoughts of suicide and has thought of at least one method but has no specific plan of action since the last visit.
Time Frame: Weeks 1, 2, 4, 6, 7, and 8, and last postbaseline observation (up to 8 weeks)
Population: The safety analysis set includes randomized participants who took 1 or more doses of study drug. This question is asked if the answer to the 'Non-Specific Active Suicidal Thoughts' question was YES, or based on the judgment of the assessor. The number analyzed includes participants with treatment assessments at the indicated time period.
Measure: Number; unit: participants
Arm/Group | Placebo | Armodafinil 150 mg/Day
Number analyzed (Participants) | 198 | 200
participants
  Week 1 (6, 5) | 1 | 1
  Week 2 (2, 6) | 0 | 0
  Week 4 (1, 7) | 0 | 0
  Week 6 (1, 3) | 0 | 0
  Week 7 (2, 2) | 0 | 0
  Week 8 (1, 3) | 0 | 0
  Endpoint (8, 12) | 1 | 0

22. Secondary Outcome: Columbia-Suicide Severity Rating Scale 'Since Last Visit' Version (C-SSRS-SLV) For Weeks 1, 2, 4, 6, 7, 8, and Endpoint For the Suicidal Ideation - Some Intent to Act Without a Specific Plan Question
Description: The C-SSRS is a clinician-rated scale that assesses suicidality from ideation to behaviors and monitors the potential emergence of suicidality in clinical studies. The C-SSRS-B (baseline) was performed at screening and the C-SSRS-SLV ('Since Last Visit') was performed at baseline and weeks 1, 2, 4, 6, 7, and 8 or last postbaseline observation.
  The Suicidal Ideation - Some Intent to Act Without a Specific Plan question records whether the participant has active suicidal thoughts of killing oneself and reports having some intent to act on such thoughts since the last visit.
Time Frame: Weeks 1, 2, 4, 6, 7, and 8, and last postbaseline observation (up to 8 weeks)
Population: as for outcome 21
Measure: Number; unit: participants
Arm/Group | Placebo | Armodafinil 150 mg/Day
Number analyzed (Participants) | 198 | 200
participants
  Week 1 (6, 5) | 0 | 0
  Week 2 (2, 6) | 0 | 0
  Week 4 (1, 7) | 0 | 0
  Week 6 (1, 3) | 0 | 0
  Week 7 (2, 2) | 0 | 0
  Week 8 (1, 3) | 0 | 0
  Endpoint (8, 12) | 0 | 0

23. Secondary Outcome: Columbia-Suicide Severity Rating Scale 'Since Last Visit' Version (C-SSRS-SLV) For Weeks 1, 2, 4, 6, 7, 8, and Endpoint For the Suicidal Ideation - Specific Plan and Intent Question
Description: The C-SSRS is a clinician-rated scale that assesses suicidality from ideation to behaviors and monitors the potential emergence of suicidality in clinical studies. The C-SSRS-B (baseline) was performed at screening and the C-SSRS-SLV ('Since Last Visit') was performed at baseline and weeks 1, 2, 4, 6, 7, and 8 or last postbaseline observation.
  The Suicidal Ideation - Specific Plan and Intent question records whether the participant has active suicidal thoughts of killing oneself with details of plan fully or partially worked out and the participant has some intent to carry out the plan since the last visit.
Time Frame: Weeks 1, 2, 4, 6, 7, and 8, and last postbaseline observation (up to 8 weeks)
Population: as for outcome 21
Measure: Number; unit: participants
Arm/Group | Placebo | Armodafinil 150 mg/Day
Number analyzed (Participants) | 198 | 200
participants
  Week 1 (6, 5) | 1 | 0
  Week 2 (2, 6) | 0 | 0
  Week 4 (1, 7) | 0 | 0
  Week 6 (1, 3) | 0 | 0
  Week 7 (2, 2) | 0 | 0
  Week 8 (1, 3) | 0 | 0
  Endpoint (8, 12) | 1 | 0

ADVERSE EVENTS:
Time Frame: Day 1 to Week 9
Arm/Group | Armodafinil 150 mg/Day | Placebo
Serious Adverse Events (participants affected / at risk) | 5/200 | 6/198
Other Adverse Events (participants affected / at risk) | 37/200 | 21/198
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Armodafinil 150 mg/Day (N=200) | Placebo (N=198)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Unintended pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Bipolar I disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Hypomania (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Social stay hospitalisation (Social circumstances) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Armodafinil 150 mg/Day (N=200) | Placebo (N=198)
Nausea (Gastrointestinal disorders) | 12 (13) | 7 (7)
Headache (Nervous system disorders) | 29 (35) | 15 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.